CLINICAL TRIAL: NCT05997641
Title: A Double-Blind, Randomized, Placebo-Controlled, First-in-Human Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Orally Administered DF-003 Following Single (Part 1) and Multiple (Part 2) Ascending Doses in Healthy Subjects
Brief Title: Evaluating the Safety, Tolerability, and Pharmacokinetics of DF-003 in Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Yao Yuan Biotechnology Ltd. (also known as Drug Farm) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DF-003-1001
Record Dates: First submitted 2023-08-01; First posted 2023-08-18 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Healthy; Safety and Tolerability
Keywords: DF-003

STUDY DESIGN:
Intervention Model Description: The study will include 2 parts: 1) Single ascending dose phase with optional food effect (FE) assessment, and 2) multiple ascending dose phase.
Who Masked: Participant, Investigator
Masking Description: Each enrolled participant will be assigned a randomization code generated with a computer program. Once generated, the randomization code will be final and will not be modified.
  The randomization code will not be available to the personnel of the bioanalytical facility until the bioanalytical phase of the study has been completed. The treatment assignment will not be known by the study participants. Furthermore, the randomization code will not be available to the physician and clinical staff involved in the collection, monitoring, revision, or evaluation of adverse events, as well as clinical staff who could have an impact on the outcome of the study.
  The preparation and/or administration of the drug products will be done by designated personnel that are not directly involved in the clinical aspects of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DF-003 (Single Ascending Dose, Part 1) (Experimental): Participants will receive a single oral dose of 3 mg DF-003 (1 mg x 3).
  Interventions: Drug: DF-003
- Placebo (Single Ascending Dose, Part 1) (Placebo Comparator): Visually matching 0 mg DF-003 capsules.
  Interventions: Drug: Placebo
- DF-003 (Multiple Ascending Doses, Part 2) (Experimental): Participants will receive DF-003 once daily by oral administration for 14 days. The specific doses given will be based on data collected in Part 1 of the study. This part of the study may include 1 mg, 5 mg, or 25 mg capsules.
  Interventions: Drug: DF-003
- Placebo (Multiple Ascending Doses, Part 2) (Placebo Comparator): Visually matching 0 mg DF-003 capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DF-003 — Oral administration by capsules (1 mg, 5 mg, or 25 mg).
  Arms: DF-003 (Multiple Ascending Doses, Part 2); DF-003 (Single Ascending Dose, Part 1)
Drug: Placebo — Visually matching 0 mg DF-003 capsules.
  Arms: Placebo (Multiple Ascending Doses, Part 2); Placebo (Single Ascending Dose, Part 1)

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, and pharmacokinetics (PK; drug metabolism) of DF-003 after oral administration of single and multiple ascending doses in healthy subjects. The choice of using healthy subjects is standard in establishing the preliminary safety and PK profile of a drug.

DF-003 is a potent small molecule inhibitor of alpha-kinase 1 (ALPK1), which plays an important role in immunity and inflammation. DF-003 can inhibit the immune inflammatory response and has been shown to reduce renal fibrosis in preclinical models. Thus, this study aims to determine the role of DF-003 in the treatment of chronic kidney disease.

This study will include 2 parts. Part 1 is a single ascending dose (SAD) phase with an optional food effect (FE) assessment, while Part 2 is a multiple ascending dose (MAD) phase. Part 1 - SAD Phase with optional FE assessment will include approximately 64 subjects (up to 8 cohorts of 8 subjects each) and Part 2 - MAD Phase will include approximately 32 subjects (up to 4 cohorts of 8 subjects each). Therefore, up to 96 subjects will be included in the study.

Study participants will be screened approximately 42 days within the first scheduled administration of study medication. Screening data will be reviewed to determine subject eligibility. In Part 1, subjects will be randomly assigned to receive a single oral dose of DF-003 (3 x 1 milligram capsules) or matching placebo. The doses to be evaluated in Part 2 will be determined based on review of the available safety and PK data from Part 1.

Subjects will be monitored for adverse events (AEs) and data will be collected for physical examination, eye examination, vital signs, 12-lead electrocardiogram (ECG), Holter monitoring, and clinical laboratory findings at various timepoints throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF).
2. Ability to understand and stated willingness to comply with all study procedures and availability for the duration of the study, and likeliness to complete the study as planned, per the Investigator's opinion.
3. Healthy adult male or female.
4. If male, meets one of the following criteria:

   1. Is able to procreate and agrees not to donate sperm from the first study drug administration to at least 90 days after the last study drug administration in addition to:

      * Having a female partner who is postmenopausal, surgically sterile, or otherwise incapable of becoming pregnant, OR
      * Having a female partner who is a woman of childbearing potential and agrees to use a highly effective method of contraception from the first study drug administration to at least 90 days after the last study drug administration, OR
   2. Is unable to procreate; defined as surgically sterile (ie, has undergone a vasectomy at least 180 days prior to the first study drug administration).
5. If female, meets one of the following criteria:

   1. Physiological postmenopausal status, defined as the following:

      * Amenorrhea for at least 12 months prior to the first study drug administration (without an alternative medical condition); AND
      * Follicle stimulating hormone (FSH) levels ≥40 mIU/mL at Screening;
      * In the absence of 12 months of amenorrhea, 2 FSH measurements at least 3 months apart and in the postmenopausal range must be documented.
   2. Surgical postmenopausal status, defined as having had a bilateral oophorectomy or bilateral salpingo-oophorectomy with FSH levels ≥ 40 mIU/mL at Screening.
6. Aged at least 18 years but not older than 55 years at the time of Screening.
7. Body mass index (BMI) within 18.0 kg/m^2 to 32.0 kg/m^2, inclusively.
8. Non- or ex-smoker (An ex-smoker is defined as someone who completed stopped using nicotine products for at least 3 months prior to the first study drug administration).
9. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination, vital signs, eye examination, and/or ECG, as determined by an Investigator.
10. A 12-lead ECG that meets the following criteria (ECG intervals will be based on the mean value of triplicate ECGs [rounded to the nearest whole number] collected at Screening):

    * Heart rate ≥45 to ≤100 beats per minute
    * QT interval corrected for heart rate (QTc) according to Fridericia's formula (QTcF) ≤450 ms (males) or ≤470 ms (females)
    * QRS interval <120 ms
    * PR interval ≤200 ms

Exclusion Criteria:

1. Female who is lactating.
2. Female who is pregnant according to the pregnancy test at Screening or prior to the first study drug administration
3. Female using the following systemic contraceptives: oral, patch or vaginal ring, in the 28 days prior to the first study drug administration.
4. Female using hormone replacement therapy in the 28 days prior to the first study drug administration.
5. Female using the following systemic contraceptives: injections or implant, or hormone-releasing intrauterine device in the 13 weeks prior to the first study drug administration.
6. History of significant hypersensitivity to products related to DF-003 (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs.
7. Presence or history of significant gastrointestinal, liver or kidney disease, or surgery (with the exception of cholecystectomy and appendectomy) that may affect drug bioavailability.
8. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic, rheumatologic, neoplastic, metabolic, or dermatologic disease.
9. Presence of clinically significant ECG abnormalities at the Screening visit, as defined by medical judgment.
10. Use of contact lenses or eyeglasses.
11. Presence of clinically significant visual acuity or slit-lamp biomicroscopy abnormalities at the Screening visit, as defined by medical judgement.
12. History or family history of chronic inflammatory skin disease (eg, psoriasis, atopic dermatitis, drug-related rash, or chronic urticaria), or immune or autoimmune related disorders, diseases, or syndromes.
13. Major surgery (eg, requiring general anesthesia) within 12 weeks before Screening, during the study, or within 12 weeks after the last dose of study drug. NOTE: Subjects with planned surgical procedures to be conducted under local anesthesia may participate.
14. Presence of renal dysfunction at Screening (eg, estimated glomerular filtration rate < 90 mL/min/1.73 m^2 calculated by the Chronic Kidney Disease Epidemiology Collaboration formula).
15. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic).
16. Any clinically significant illness including current acute or chronic infections in the 28 days prior to the first study drug administration.
17. Use of any prescription drugs in the 28 days prior to the first study drug administration, that in the opinion of an Investigator would put into question the status of the participant as healthy.
18. Use of St. John's wort in the 28 days prior to the first study drug administration.
19. Use of any over-the-counter medications 7 days prior to the first study drug administration. Subjects will be reminded that over-the-counter medications include cold preparations, aspirin, vitamins and natural products used for therapeutic benefits, and antacid preparations.
20. Positive test result for alcohol and/or drugs of abuse at Screening or prior to the first drug administration.
21. Positive screening results to HIV Ag/Ab combo, hepatitis B surface antigen, or hepatitis C virus tests.
22. Any other clinically significant abnormalities in laboratory test results at Screening that would, in the opinion of an Investigator, increase the subject's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data.
23. Intake of an IP in the 4 weeks (or 5 half-lives, whichever is longer) prior to the first study drug administration.
24. Intake of any biological products in the 12 months prior to the first study drug administration.
25. Current participation in another clinical or medical interventional research study.
26. Employee of the Sponsor, Investigator or study site with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, as well as family members of the employees or Investigator.
27. Donation of plasma in the 7 days prior to the first study drug administration.
28. Donation of 1 unit of blood to American Red Cross or equivalent organization or donation of over 500 mL of blood in the 56 days prior to the first study drug administration.
29. Presence or history of eye lens opacification (cataracts) and eye lens degeneration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-03-23 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 83 days
  Safety and Tolerability
Incidence of Serious Adverse Events (SAEs) | Up to 83 days
  Safety and Tolerability

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) for DF-003 | Up to 83 days
  Pharmacokinetics
Time to maximum plasma concentration (tmax) for DF-003 | Up to 83 days
  Pharmacokinetics
Area under the plasma concentration-time curve from zero to the time of the last quantifiable concentration (AUC(0-t)) for DF-003 | Up to 83 days
  Pharmacokinetics
Area under the plasma concentration-time curve from zero to infinity ((AUC(0-∞)) for DF-003 | Up to 83 days
  Pharmacokinetics
Terminal half-life (t½) for DF-003 | Up to 83 days
  Pharmacokinetics
Apparent plasma clearance of drug after extravascular administration (CL/F) for DF-003 | Up to 83 days
  Pharmacokinetics
Apparent volume of distribution after extravascular administration (Vz/F) for DF-003 | Up to 83 days
  Pharmacokinetics
Maximum plasma concentration at steady state (Cmax,ss) for DF-003 | Up to 83 days
  Pharmacokinetics
Time to steady state Cmax (Tss,max) for DF-003 | Up to 83 days
  Pharmacokinetics
Concentration at time t (Ct) for DF-003 | Up to 83 days
  Pharmacokinetics
Concentration immediately before next dose (Ctrough) for DF-003 | Up to 83 days
  Pharmacokinetics
Apparent plasma clearance of drug after extravascular administration at steady state (CLss/F) for DF-003 | Up to 83 days
  Pharmacokinetics
Apparent volume of distribution at steady state after extravascular administration (Vz,ss/F) for DF-003 | Up to 83 days
  Pharmacokinetics
Accumulation ratio (Rac) at Cmax for DF-003 | Up to 83 days
  Pharmacokinetics
Accumulation ratio area under the concentration-time curve for DF-003 | Up to 83 days
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Javid Ghandehari, MD, Principal Investigator — Interventional Pain Management Physician Anesthesiologist, Altasciences
Locations (1):
- Altasciences Clinical Los Angeles, Inc, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hallan SI, Ovrehus MA, Romundstad S, Rifkin D, Langhammer A, Stevens PE, Ix JH. Long-term trends in the prevalence of chronic kidney disease and the influence of cardiovascular risk factors in Norway. Kidney Int. 2016 Sep;90(3):665-73. doi: 10.1016/j.kint.2016.04.012. Epub 2016 Jun 22. PMID 27344204
- [Background] Murphy D, McCulloch CE, Lin F, Banerjee T, Bragg-Gresham JL, Eberhardt MS, Morgenstern H, Pavkov ME, Saran R, Powe NR, Hsu CY; Centers for Disease Control and Prevention Chronic Kidney Disease Surveillance Team. Trends in Prevalence of Chronic Kidney Disease in the United States. Ann Intern Med. 2016 Oct 4;165(7):473-481. doi: 10.7326/M16-0273. Epub 2016 Aug 2. PMID 27479614
- [Background] Shin HY, Kang HT. Recent trends in the prevalence of chronic kidney disease in Korean adults: Korean National Health and Nutrition Examination Survey from 1998 to 2013. J Nephrol. 2016 Dec;29(6):799-807. doi: 10.1007/s40620-016-0280-y. Epub 2016 Mar 4. PMID 26943182
- [Background] Decleves AE, Sharma K. Novel targets of antifibrotic and anti-inflammatory treatment in CKD. Nat Rev Nephrol. 2014 May;10(5):257-67. doi: 10.1038/nrneph.2014.31. Epub 2014 Mar 25. PMID 24662433
- [Background] Jha V, Garcia-Garcia G, Iseki K, Li Z, Naicker S, Plattner B, Saran R, Wang AY, Yang CW. Chronic kidney disease: global dimension and perspectives. Lancet. 2013 Jul 20;382(9888):260-72. doi: 10.1016/S0140-6736(13)60687-X. Epub 2013 May 31. PMID 23727169
- [Background] Lopez-Novoa JM, Martinez-Salgado C, Rodriguez-Pena AB, Lopez-Hernandez FJ. Common pathophysiological mechanisms of chronic kidney disease: therapeutic perspectives. Pharmacol Ther. 2010 Oct;128(1):61-81. doi: 10.1016/j.pharmthera.2010.05.006. Epub 2010 Jun 19. PMID 20600306
- [Background] Khwaja A, El Kossi M, Floege J, El Nahas M. The management of CKD: a look into the future. Kidney Int. 2007 Dec;72(11):1316-23. doi: 10.1038/sj.ki.5002489. Epub 2007 Aug 15. PMID 17700639
- [Background] Liu Y. Cellular and molecular mechanisms of renal fibrosis. Nat Rev Nephrol. 2011 Oct 18;7(12):684-96. doi: 10.1038/nrneph.2011.149. PMID 22009250
- [Background] Yu J, Mao S, Zhang Y, Gong W, Jia Z, Huang S, Zhang A. MnTBAP Therapy Attenuates Renal Fibrosis in Mice with 5/6 Nephrectomy. Oxid Med Cell Longev. 2016;2016:7496930. doi: 10.1155/2016/7496930. Epub 2016 Feb 17. PMID 26989454
- [Background] Humphreys BD. Mechanisms of Renal Fibrosis. Annu Rev Physiol. 2018 Feb 10;80:309-326. doi: 10.1146/annurev-physiol-022516-034227. Epub 2017 Oct 25. PMID 29068765
- [Background] Kefaloyianni E, Muthu ML, Kaeppler J, Sun X, Sabbisetti V, Chalaris A, Rose-John S, Wong E, Sagi I, Waikar SS, Rennke H, Humphreys BD, Bonventre JV, Herrlich A. ADAM17 substrate release in proximal tubule drives kidney fibrosis. JCI Insight. 2016 Aug 18;1(13):e87023. doi: 10.1172/jci.insight.87023. PMID 27642633
- [Background] Levey AS, Atkins R, Coresh J, Cohen EP, Collins AJ, Eckardt KU, Nahas ME, Jaber BL, Jadoul M, Levin A, Powe NR, Rossert J, Wheeler DC, Lameire N, Eknoyan G. Chronic kidney disease as a global public health problem: approaches and initiatives - a position statement from Kidney Disease Improving Global Outcomes. Kidney Int. 2007 Aug;72(3):247-59. doi: 10.1038/sj.ki.5002343. Epub 2007 Jun 13. PMID 17568785
- [Background] Anders HJ, Belemezova E, Eis V, Segerer S, Vielhauer V, Perez de Lema G, Kretzler M, Cohen CD, Frink M, Horuk R, Hudkins KL, Alpers CE, Mampaso F, Schlondorff D. Late onset of treatment with a chemokine receptor CCR1 antagonist prevents progression of lupus nephritis in MRL-Fas(lpr) mice. J Am Soc Nephrol. 2004 Jun;15(6):1504-13. doi: 10.1097/01.asn.0000130082.67775.60. PMID 15153561
- [Background] Duffield JS. Cellular and molecular mechanisms in kidney fibrosis. J Clin Invest. 2014 Jun;124(6):2299-306. doi: 10.1172/JCI72267. Epub 2014 Jun 2. PMID 24892703
- [Background] Kurts C, Panzer U, Anders HJ, Rees AJ. The immune system and kidney disease: basic concepts and clinical implications. Nat Rev Immunol. 2013 Oct;13(10):738-53. doi: 10.1038/nri3523. Epub 2013 Sep 16. PMID 24037418
- [Background] Lopez-de la Mora DA, Sanchez-Roque C, Montoya-Buelna M, Sanchez-Enriquez S, Lucano-Landeros S, Macias-Barragan J, Armendariz-Borunda J. Role and New Insights of Pirfenidone in Fibrotic Diseases. Int J Med Sci. 2015 Oct 14;12(11):840-7. doi: 10.7150/ijms.11579. eCollection 2015. PMID 26640402
- [Background] Tampe D, Zeisberg M. Potential approaches to reverse or repair renal fibrosis. Nat Rev Nephrol. 2014 Apr;10(4):226-37. doi: 10.1038/nrneph.2014.14. Epub 2014 Feb 11. PMID 24514753
- [Background] Wang SN, LaPage J, Hirschberg R. Role of glomerular ultrafiltration of growth factors in progressive interstitial fibrosis in diabetic nephropathy. Kidney Int. 2000 Mar;57(3):1002-14. doi: 10.1046/j.1523-1755.2000.00928.x. PMID 10720953
- [Background] Lee SY, Kim SI, Choi ME. Therapeutic targets for treating fibrotic kidney diseases. Transl Res. 2015 Apr;165(4):512-30. doi: 10.1016/j.trsl.2014.07.010. Epub 2014 Aug 13. PMID 25176603
- [Background] Chow FY, Nikolic-Paterson DJ, Ma FY, Ozols E, Rollins BJ, Tesch GH. Monocyte chemoattractant protein-1-induced tissue inflammation is critical for the development of renal injury but not type 2 diabetes in obese db/db mice. Diabetologia. 2007 Feb;50(2):471-80. doi: 10.1007/s00125-006-0497-8. Epub 2006 Dec 12. PMID 17160673
- [Background] Kanamori H, Matsubara T, Mima A, Sumi E, Nagai K, Takahashi T, Abe H, Iehara N, Fukatsu A, Okamoto H, Kita T, Doi T, Arai H. Inhibition of MCP-1/CCR2 pathway ameliorates the development of diabetic nephropathy. Biochem Biophys Res Commun. 2007 Sep 7;360(4):772-7. doi: 10.1016/j.bbrc.2007.06.148. Epub 2007 Jul 6. PMID 17631861
- [Background] Kang YS, Lee MH, Song HK, Ko GJ, Kwon OS, Lim TK, Kim SH, Han SY, Han KH, Lee JE, Han JY, Kim HK, Cha DR. CCR2 antagonism improves insulin resistance, lipid metabolism, and diabetic nephropathy in type 2 diabetic mice. Kidney Int. 2010 Nov;78(9):883-94. doi: 10.1038/ki.2010.263. Epub 2010 Aug 4. PMID 20686445
- [Background] Kitagawa K, Wada T, Furuichi K, Hashimoto H, Ishiwata Y, Asano M, Takeya M, Kuziel WA, Matsushima K, Mukaida N, Yokoyama H. Blockade of CCR2 ameliorates progressive fibrosis in kidney. Am J Pathol. 2004 Jul;165(1):237-46. doi: 10.1016/S0002-9440(10)63292-0. PMID 15215179
- [Background] Sullivan T, Miao Z, Dairaghi DJ, Krasinski A, Wang Y, Zhao BN, Baumgart T, Ertl LS, Pennell A, Seitz L, Powers J, Zhao R, Ungashe S, Wei Z, Boring L, Tsou CL, Charo I, Berahovich RD, Schall TJ, Jaen JC. CCR2 antagonist CCX140-B provides renal and glycemic benefits in diabetic transgenic human CCR2 knockin mice. Am J Physiol Renal Physiol. 2013 Nov 1;305(9):F1288-97. doi: 10.1152/ajprenal.00316.2013. Epub 2013 Aug 28. PMID 23986513
- [Background] Poveda J, Tabara LC, Fernandez-Fernandez B, Martin-Cleary C, Sanz AB, Selgas R, Ortiz A, Sanchez-Nino MD. TWEAK/Fn14 and Non-Canonical NF-kappaB Signaling in Kidney Disease. Front Immunol. 2013 Dec 10;4:447. doi: 10.3389/fimmu.2013.00447. PMID 24339827
- [Background] Volpini RA, Costa RS, da Silva CG, Coimbra TM. Inhibition of nuclear factor-kappaB activation attenuates tubulointerstitial nephritis induced by gentamicin. Nephron Physiol. 2004;98(4):p97-106. doi: 10.1159/000081558. PMID 15627798
- [Background] Ding W, Yang L, Zhang M, Gu Y. Chronic inhibition of nuclear factor kappa B attenuates aldosterone/salt-induced renal injury. Life Sci. 2012 Apr 20;90(15-16):600-6. doi: 10.1016/j.lfs.2012.02.022. Epub 2012 Mar 3. PMID 22406301
- [Background] Horii Y, Muraguchi A, Iwano M, Matsuda T, Hirayama T, Yamada H, Fujii Y, Dohi K, Ishikawa H, Ohmoto Y, et al. Involvement of IL-6 in mesangial proliferative glomerulonephritis. J Immunol. 1989 Dec 15;143(12):3949-55. PMID 2592764
- [Background] Fattori E, Cappelletti M, Costa P, Sellitto C, Cantoni L, Carelli M, Faggioni R, Fantuzzi G, Ghezzi P, Poli V. Defective inflammatory response in interleukin 6-deficient mice. J Exp Med. 1994 Oct 1;180(4):1243-50. doi: 10.1084/jem.180.4.1243. PMID 7931061
- [Background] Liang B, Gardner DB, Griswold DE, Bugelski PJ, Song XY. Anti-interleukin-6 monoclonal antibody inhibits autoimmune responses in a murine model of systemic lupus erythematosus. Immunology. 2006 Nov;119(3):296-305. doi: 10.1111/j.1365-2567.2006.02433.x. PMID 17067309
- [Background] Jones SA, Fraser DJ, Fielding CA, Jones GW. Interleukin-6 in renal disease and therapy. Nephrol Dial Transplant. 2015 Apr;30(4):564-74. doi: 10.1093/ndt/gfu233. Epub 2014 Jul 10. PMID 25011387
- [Background] Zhou P, She Y, Dong N, Li P, He H, Borio A, Wu Q, Lu S, Ding X, Cao Y, Xu Y, Gao W, Dong M, Ding J, Wang DC, Zamyatina A, Shao F. Alpha-kinase 1 is a cytosolic innate immune receptor for bacterial ADP-heptose. Nature. 2018 Sep;561(7721):122-126. doi: 10.1038/s41586-018-0433-3. Epub 2018 Aug 15. PMID 30111836
- [Background] Matoba K, Takeda Y, Nagai Y, Kawanami D, Utsunomiya K, Nishimura R. Unraveling the Role of Inflammation in the Pathogenesis of Diabetic Kidney Disease. Int J Mol Sci. 2019 Jul 10;20(14):3393. doi: 10.3390/ijms20143393. PMID 31295940
- [Background] Yamada Y, Nishida T, Ichihara S, Kato K, Fujimaki T, Oguri M, Horibe H, Yoshida T, Watanabe S, Satoh K, Aoyagi Y, Fukuda M, Sawabe M. Identification of chromosome 3q28 and ALPK1 as susceptibility loci for chronic kidney disease in Japanese individuals by a genome-wide association study. J Med Genet. 2013 Jun;50(6):410-8. doi: 10.1136/jmedgenet-2013-101518. Epub 2013 Mar 28. PMID 23539754
- [Background] Shimokata S, Oguri M, Fujimaki T, Horibe H, Kato K, Yamada Y. Association between polymorphisms of the alpha-kinase 1 gene and type 2 diabetes mellitus in community-dwelling individuals. Biomed Rep. 2013 Nov;1(6):940-944. doi: 10.3892/br.2013.173. Epub 2013 Sep 25. PMID 24649057
- [Background] Fujimaki T, Horibe H, Oguri M, Kato K, Yamada Y. Association of genetic variants of the alpha-kinase 1 gene with myocardial infarction in community-dwelling individuals. Biomed Rep. 2014 Jan;2(1):127-131. doi: 10.3892/br.2013.190. Epub 2013 Oct 30. PMID 24649083
- [Background] Yamada Y, Matsui K, Takeuchi I, Fujimaki T. Association of genetic variants with coronary artery disease and ischemic stroke in a longitudinal population-based genetic epidemiological study. Biomed Rep. 2015 May;3(3):413-419. doi: 10.3892/br.2015.440. Epub 2015 Mar 2. PMID 26137247
- [Background] Yamada Y, Matsui K, Takeuchi I, Fujimaki T. Association of genetic variants with dyslipidemia and chronic kidney disease in a longitudinal population-based genetic epidemiological study. Int J Mol Med. 2015 May;35(5):1290-300. doi: 10.3892/ijmm.2015.2152. Epub 2015 Mar 20. PMID 25813695
- [Background] Yamada Y, Matsui K, Takeuchi I, Oguri M, Fujimaki T. Association of genetic variants of the alpha-kinase 1 gene with type 2 diabetes mellitus in a longitudinal population-based genetic epidemiological study. Biomed Rep. 2015 May;3(3):347-354. doi: 10.3892/br.2015.439. Epub 2015 Mar 2. PMID 26137234